CLINICAL TRIAL: NCT05068102
Title: An Open Label Phase I PET Imaging Study to Investigate the Bio-distribution and Tumor Uptake of [89Zr]Zr-BI 765063 and [89Zr]Zr-BI 770371 in Patients With Head and Neck Squamous Cell Carcinoma, Non-small Cell Lung Cancer or Melanoma Who Are Treated With Ezabenlimab
Brief Title: A Study to Test How BI 765063 and BI 770371 Are Taken up in Tumours of People With Different Types of Advanced Cancer Who Are Also Taking Ezabenlimab
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1443-0003; 2021-001063-25 (EudraCT Number)
Record Dates: First submitted 2021-09-19; First posted 2021-10-05 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck (HNSCC); Melanoma; Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma; Squamous Cell Carcinoma of Head and Neck; Melanoma; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: The trial is divided in 2 parts:
  In Part 1 of each arm, the patients will be entered sequentially. After review of Part 1 data for each arm, the Data Review Committee (DRC) will make the decision whether or not to initiate Part 2 for each arm.
  Patients entered in Part 2 will be treated in various dose cohorts of BI 765063 (Arm A) or BI 770371 (Arm B) at Cycle 2 and these dose cohorts will be managed sequentially based on the DRC decision.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: BI 765063; Drug: Ezabenlimab; Drug: [89Zr]Zr- BI 765063
- Arm B (Experimental)
  Interventions: Drug: Ezabenlimab; Drug: BI 770371; Drug: [89Zr]Zr- BI 770371

INTERVENTIONS:
Drug: BI 765063 — BI 765063
  Arms: Arm A
Drug: Ezabenlimab — Ezabenlimab
Drug: [89Zr]Zr- BI 765063 — [89Zr]Zr- BI 765063, specifically radiolabelled for immune-Positron Emission Tomography (PET)
  Arms: Arm A
Drug: BI 770371 — BI 770371
  Arms: Arm B
Drug: [89Zr]Zr- BI 770371 — [89Zr]Zr- BI 770371, specifically radiolabelled for immune-PET
  Arms: Arm B

SUMMARY:
This study is open to adults with advanced head and neck cancer, skin cancer, or non-small cell lung cancer. People can take part if previous treatments were not successful.

The purpose of this study is to find out how 2 medicines called BI 765063 and BI 770371 are taken up in the tumours and how they get distributed in the body. In addition to BI 765063 or BI 770371, participants also receive ezabenlimab. BI 765063, BI 770371 and ezabenlimab are antibodies that may help the immune system fight cancer. Such therapies are also called immune checkpoint inhibitors.

Participants get either BI 765063 or BI 770371 in combination with ezabenlimab as an infusion into a vein every 3 weeks. In the first weeks, doctors check how BI 765063 and BI 770371 are taken up in tumours. To do so, the doctors use imaging methods (PET/CT scans). For this, participants get BI 765063 or BI 770371 injected in a labelled form up to 2 times.

Participants can stay in the study as long as they benefit from treatment and can tolerate it. The doctors regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria:

* Signed and dated, written informed consent form (ICF) prior to any trial-specific procedures
* Male or female aged ≥ 18 years (no upper limit of age) at the time of ICF signature
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of at least 3 months
* For Arm A, only patients with a Signal Regulatory Protein-alpha (SIRPα) polymorphism V1/V1 will be eligible; SIRPα polymorphism will be assessed in blood sampling (patient deoxyribonucleic acid (DNA)) in a central laboratory; V1 allele is understood to include V1 and potential V1-like alleles. If, at a later time, V1/V2 heterozygous patients are considered for inclusion in this Arm of the trial, these patients will require to be centrally confirmed with at least one V1 allele.
* Patients with histologically or cytologically documented advanced/metastatic primary or recurrent Head and Neck Squamous Cell Carcinoma (HNSCC), melanoma, Non-Small Cell Lung Cancer (NSCLC) who failed or are not eligible to standard therapy
* Patients with at least one measurable lesion are allowed as per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1
* Patient must have at least one Positron Emission Tomography (PET) imageable and evaluable tumor lesion with a diameter of at least 20 millimeter Further inclusion criteria apply.

Exclusion criteria:

* Patients with symptomatic/active central nervous system (CNS) metastases; patients with previously treated brain metastases are eligible if there is no evidence of progression for at least 28 days before the first study treatment administration, as ascertained by clinical examination and brain imaging (Magnetic Resonance Imaging (MRI) or Computed Tomography (CT)) during the screening period
* Other tumor location necessitating an urgent therapeutic intervention (e.g., palliative care, surgery or radiation therapy, such as spinal cord compression, other compressive mass, uncontrolled painful lesion, bone fracture)
* Presence of other active invasive cancers other than the one treated in this trial within 5 years prior to screening (or less, pending discussion with sponsor), except appropriately treated basal cell carcinoma of the skin, or in situ carcinoma of uterine cervix, or other local tumors considered cured by local treatment
* Patients with active autoimmune disease or a documented history of autoimmune disease, that requires systemic treatment (i.e. corticosteroids or immunosuppressive drugs); except patients with vitiligo, resolved childhood asthma/atopy, alopecia, or any chronic skin condition that does not require systemic therapy, patients with autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone and/or controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible
* Known severe infusion related reactions to monoclonal antibodies (Grade ≥ 3 National Cancer Institute (NCI)- Common Terminology Criteria for Adverse Events (CTCAE) v5.0) and patients removed from previous anti-Programmed-cell-death-protein-1 (PD-1) or anti-Programmed-cell-death ligand-1 (PD-L1) therapy because of a severe or life-threatening immune-related adverse event (irAE) (Grade ≥ 3 NCI-CTCAE v5.0)
* Patients receiving systemic treatment with any immunosuppressive medication within one-week prior to treatment start with SIRPα antibody (BI 765063 or BI 770371) and ezabenlimab; steroids of max. 10 mg prednisolone equivalent per day are allowed, topical and inhaled steroids are not considered as immunosuppressive
* Patients who have interstitial lung disease or active, non-infectious pneumonitis.
* Patients with uncontrolled disease-related metabolic disorders (e.g., hypercalcemia, Syndrome of Inappropriate of AntiDiuretic Hormone Secretion (SIADH)) or uncontrolled diabetes Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2026-04-03 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Arm A: Relative change from baseline (Cycle 1, up to Day 7) of peak Standardized Uptake Values (SUVs) of [89Zr]Zr-BI 765063 in up to five target lesions at post BI 765063 treatment scanning time points (Cycle 2, up to Day 7) | up to 33 months
  peak SUVs are measured via Positron Emission Tomography (PET) scan
Arm B: Relative change from baseline (Cycle 1, up to Day 7) of peak Standardized Uptake Values (SUVs) of [89Zr]Zr-BI 770371 in up to five target lesions at post BI 770371 treatment scanning time points (Cycle 2, up to Day 7) | up to 33 months
  peak SUVs are measured via Positron Emission Tomography (PET) scan

CONTACTS AND LOCATIONS:
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com